CLINICAL TRIAL: NCT02317185
Title: CLINICAL EVALUATION OF GENEX® DS IN INSTRUMENTED POSTEROLATERAL FUSION
Status: Terminated | Type: Observational
Why Stopped: For business reasons / product no longer available from Sponsor
Sponsor: Spine Wave (Industry)
Responsible Party: Sponsor
Other Study IDs: GEN-1401
Record Dates: First submitted 2014-12-08; First posted 2014-12-15 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Stenosis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Constriction, Pathologic | interventions — Bone Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: genex bone graft with bone graft
Other: autogenous bone graft

SUMMARY:
The overall goal of this clinical study is to characterize the fusion rate of geneX® ds bone graft substitute in comparison to autograft, which is considered the gold standard for posterolateral fusion. Assessments are made using AP and Lateral x-rays, F/E x-rays, and CT scans geneX® ds has been cleared by the FDA for use in these procedures; however this study will allow more detailed characterization of geneX® ds performance in the long-term (1 year). By using the patient as their own control, direct comparison to autograft can be performed while minimizing other variables.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18-75 years of age
* Have ability to understand the requirements of the study, to provide written informed consent, and to comply with the study protocol
* Have a spinal condition of the lumbar spine (L1-S1) requiring instrumented posterolateral fusion at one or two levels

Exclusion Criteria:

* Patients undergoing instrumented fusion for trauma, tumor, psuedoarthrosis, or same- - level recurrent stenosis
* Patients where placing graft material on both sides (posterolateral gutters) is not possible, for example in the case of a complete facetectomy
* Patients requiring instrumented fusion in the cervical or thoracic spine
* Extraspinal cause of back pain such as trauma, infection, instrumentation failure, or neoplasm
* Severe degenerative bone disease
* Hypercalcemia
* Active local or systemic infection
* Morbid obesity defined as BMI > 40
* Patients who are pregnant / able to become pregnant and not following a reliable contraceptive method
* Uncooperative patients who can't or won't follow post-operative instructions including individuals who abuse drugs or alcohol
* Anatomy or other factors that prohibit safe surgical access to the surgical site
* Allergy or sensitivity to any component of the treatment procedure
* Inadequate tissue coverage over the operative site
* Inadequate bone stock or bone quality
* Fever or leukocytosis
* Uncorrectable coagulopathy or hemorrhagic diathesis
* Uncontrolled diabetes
* Severe vascular disease or cardiopulmonary conditions that present prohibitive anesthesia risk
* Neuromuscular disease or disorder
* Mental illness
* Has an active workman's compensation lawsuit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population will include adult (skeletally mature) men and women with spinal conditions for which instrumented posterolateral fusion (PLF) has been indicated as a course of treatment. Such spinal conditions may include symptomatic degenerative disc disease, spondylolisthesis (Grade I or II), or lumbar stenosis. The study is limited to those patients requiring instrumented PLF at one or two levels only. Subjects who are undergoing other spinal procedures during the same surgery (such as interbody fusions) are also eligible.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Fusion | 1 year
  Fusion will be assessed by a single, independent radiologist using study required x-rays (AP, Lateral, Flexion-Extension) and CT scans. On xray, fusion will be graded for bridging bone and lucencies. Flexion extension x-rays will also be evaluated to determine translational and angular motion. For these evaluations, fusion is defined as translational motion < 3mm and angular motion < 5º.CT assessments of fusion will include qualitative evaluation of the continuity of trabecular bone between the transverse processes, cortication at the peripheral edges of the fusion masses, and the absence of identifiable radiographic clefts. Quantitative volumetric measurements of the fusion mass will be performed by outlining the fusion area in each cross-sectional slice and summing all slices.

SECONDARY OUTCOMES:
Complications | 1 year
  Complications will be assessed by evaluating all reported adverse events. The analysis will be descriptive only.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hospital for Special Surgery, New York, New York
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina